CLINICAL TRIAL: NCT07322146
Title: Comparing Two Durations of Antibiotic Treatment for Children Hospitalized With Common Infections
Brief Title: Trial of Reducing Inpatient Antibiotic Durations in Children
Acronym: TRIAD
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 25-45723
Record Dates: First submitted 2026-01-05; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Pneumonia; Skin and Soft Tissue (SST) Infection; Urinary Tract Infections (UTIs)
Keywords: Randomized Control Trial; Double-Blinded; Antibiotic duration; Hospital Medicine; Pediatrics
MeSH Terms: conditions — Pneumonia; Infections; Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 5-day duration treatment strategy (Experimental): Participants will use the antibiotic prescribed by thier hospital care team for the first 5 days of antibiotic therapy. They will change to study medication, a placebo, for days 6-10 of therapy.
  Interventions: Drug: Study Drug Placebo
- 10-day duration treatment strategy (No Intervention): Participants will use the antibiotic prescribed by thier hospital care team for the first 5 days of antibiotic therapy. They will change to study medication, a continuation of that antibiotic, for days 6-10 of therapy.

INTERVENTIONS:
Drug: Study Drug Placebo — Placebo, medically nonactive drug
  Arms: 5-day duration treatment strategy

SUMMARY:
Infections like pneumonia, skin and soft tissue infection (also called SSTI or cellulitis), and urinary tract infections (UTI) are some of the most common reasons children get admitted to the hospital. All three of these conditions require antibiotics for treatment. Although antibiotics are needed to treat the infection and help children feel better, taking them longer than needed can negatively impact children and their families. Negative impacts include things like the burdens of taking more medications and medication side effects. There are guidelines (instructions) from expert medical organizations that suggest the number of days children need antibiotics, but they give a wide range (between 5 and 14 days). Unfortunately, these guidelines are not based on high-quality studies. National data suggests that doctors often choose on the higher end of this range when writing prescriptions for children in the hospital.

Our three caregiver co-investigators, other parents of hospitalized children, doctors, other care providers, and researchers, all believe that additional study is needed to determine the best length of antibiotic treatment that weighs both the benefits and harms of antibiotics.

The goal of our study is to understand if 5 total days of antibiotic treatment compared to 10 total days of antibiotic treatment is better for children who have been in the hospital for pneumonia, SSTI, or UTI. We will study this question through a randomized control trial. In other words, half of the children will receive 5-days of antibiotics and the other half will receive 10-days of antibiotics. Children in this study (and their caregivers) will not know how many days of antibiotics they will receive to cure their infection because some children will take a placebo (or a pill without antibiotics in it). Only the pharmacy will know if a child is getting antibiotic or placebo (for days 6-10 of treatment).

During the first phase of the trial (feasibility phase), 4 hospitals will enroll children in the study. We plan on enrolling 50 patients during this phase. We are starting with just 4 hospitals, so our study team can create and update our study plans if needed. We will closely review information about how many patients and families agree to participate, and if they have any trouble completing any part of the study. We will also interview families to understand the choice to participate in the study, the choice not to participate in the study, and what it is like to be in the study.

During the second study phase, we will enroll 1150 more patients across all 11 hospitals. Families will complete short, daily surveys until the 15th day after they started antibiotics, then a larger survey at day 15, at day 20, and at day 30. These surveys will ask about the child's symptoms and recovery from their illness, how the antibiotics are making them feel, and if they had to go back to their doctor, emergency room, or hospital. The answers to these questions will be combined to measure how well the child did, balancing feeling better and having bad effects from the antibiotics.

We will use mathematical tests to determine which antibiotic duration is better for treating these illnesses. We will complete other mathematical tests to see if all children should receive the same length of antibiotics or if certain children should be prescribed shorter courses and others longer courses.

ELIGIBILITY:
Inclusion Criteria:

We will include children and adolescents ages 60 days to 17 years and 10 months admitted to the hospital medicine service with a primary diagnosis of PNA, SSTI, or UTI receiving an antibiotic agent that is concordant with any microbiologic results and guideline-concordant. Children are eligible if they are prescribed a post-discharge antibiotic for home that is within our trial formulary.

For PNA, children must have radiographic evidence of pneumonia as read by a radiologist, and clinical diagnosis of pneumonia, and clinician prescription of guideline-concordant antibiotics for pneumonia. For SSTI, we will include children with cellulitis alone or cellulitis with abscess that was either drained or deemed too small for drainage. For UTI, children must meet guideline-specified diagnostic criteria.

Exclusion Criteria:

We will exclude any patients who live independently (without a parent or guardian in the home), including those in county or state custody. We will exclude patients who previously enrolled (i.e., consented and randomized) in the study. We will exclude patients who are not discharging home from hospital medicine service.

For all conditions, we will exclude children who require inpatient antibiotics longer than 4 days, as guidelines indicate that a child should be clinically improving to be a candidate for short duration treatment strategy. We will also exclude children discharged with >1 systemic antibiotic prescription, as this may indicate greater severity of infection or greater diagnostic uncertainty. Other exclusion criteria are also all aligned with guidelines, which exclude children that may require longer duration antibiotics or have higher risk of infections with resistant or atypical organisms, including exclusion of patients requiring >24 hours in intensive care, patients with immunodeficiency, patients who have been hospitalized in the preceding 30 days before the index hospitalization, patients who are admitted after completing more than 48 hours of outpatient antibiotics to treat the current infection, known pregnant patients, anyone who has an allergy to any of the components of the placebo, and anyone with clear alternate diagnosis, need for treatment of a concomitant diagnosis requiring antibiotics, or uncertainty regarding the qualifying diagnosis (PNA, SSTI, UTI).

For pneumonia, we will exclude children with a parapneumonic effusion larger than "trace" or "small" (based on radiologist impression), tracheostomy, high intensity neurologic impairment, cystic fibrosis, sickle cell disease, chronic respiratory failure, or received 3 or more doses of azithromycin. For SSTI, we will exclude children with surgical site infections, cellulitis around a medical device, bone or joint infections, infectious myositis or pyomyositis, implanted hardware or other deep infections, have concomitant HSV, significant chronic dermatologic conditions other than eczema, or pre-septal or orbital cellulitis. Dental abscess without overlying facial cellulitis will also be excluded. We will exclude those discharged from the hospital with a drain in place. However, any abscess at the skin would qualify even if it is drained by a subspecialist, unless it connects with an internal cavity. For UTI, we will exclude children with major genitourinary anomalies, high-grade vesicoureteral reflux, history of urologic surgery other than circumcision, indwelling urinary catheters, need for regular intermittent catheterization, or current renal abscess.

Ages: 60 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1200 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2031-08 (Estimated); Study Completion 2031-08 (Estimated)

PRIMARY OUTCOMES:
DOOR-RADAR composite outcome at day 15 | Day 15 after antibiotic initiation
  This is a composite, ordinal outcome captured through caregiver survey on day 15 after antibiotic initiation. This outcome includes 3 domains: clinical treatment failure, symptom and function recovery, and antibiotic-associated adverse effects. Each participant is assigned an ordinal outcome category (eight possible categories, each representing a unique combination of the three domains).

CONTACTS AND LOCATIONS:
Overall Officials: Sunitha V Kaiser, MD, MSc, Principal Investigator — University of California, San Francisco
Locations (10):
- United States (10):
  - Children's of Alabama, Birmingham, Alabama
  - Children's Hospital of Colorado, Aurora, Colorado
  - Children's National Hospital, Washington D.C., District of Columbia
  - Cincinnati Children's Hospital Medical Center Liberty Campus, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center-Burnet Campus, Cincinnati, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Monroe Carrell Jr Children's Hospital at Vanderbilt University Medical Center, Nashville, Tennessee
  - Primary Children's Hospital, Lehi, Utah
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Limited Data Set versions will be distributed to external collaborators with a data use agreement. Any collaborator requiring identifying data elements outside the bounds of a Limited Data Set will first be added formally as research personnel. The Data Coordinatin Center will preserve research data and documentation for sharing and reuse, for 7 years after the study's final report.
Supporting Information: Study Protocol, SAP, ICF, CSR